CLINICAL TRIAL: NCT03496480
Title: Stroke complicAtions After TraUmatic expeRieNces and Stress - a Retrospective Cohort Study
Brief Title: Stroke complicAtions After TraUmatic expeRieNces and Stress
Acronym: SATURN
Status: Completed | Type: Observational
Sponsor: Johanna Schöner (Other)
Responsible Party: Sponsor-Investigator, Johanna Schöner, study doctor, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: EA2/113/16
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Stroke
Keywords: ptsd; stress; traumatization
MeSH Terms: conditions — Stroke; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Questionnaires — Psychological questionnaires: BTQ, IES-R, 7-items-short Screening scale, BDI, SF-36

SUMMARY:
The primary aim of this retrospective cohort study is to test the hypothesis that previous traumatization (long) before an ischemic stroke increases the degree of stroke-induced PTSD symptoms at 9-13 months after the stroke event. Secondary outcome parameters include quality of life and depression.

DETAILED DESCRIPTION:
Neuropsychiatric consequences of brain ischemia play a critical role in shaping long-term stroke outcome. Unfortunately, however, as of now, clinical research and clinical practice have not adequately addressed this growing challenge. A good case in point is posttraumatic stress disorder (PTSD). Previous trauma exposure and posttraumatic stress symptoms may increase the risk of cardiovascular events (Sumner et al., 2015). Moreover, unbeknownst to most clinical neurologists, a significant portion (approximately 25%) of their stroke patients develop symptoms of post-traumatic stress disorder (PTSD) within the first year post-event. PTSD-related symptoms after an acute coronary syndrome increase the risk of recurrent cardiac events and mortality (Edmondson et al., 2012). Similarly, stroke-induced PTSD has been linked with worse long term stroke outcome, in particular, recurrent stroke, greater disability, non-adherence to medications, and comorbidities (Goldfinger et al., 2014; Kronish et al., 2012).

For a period of 22 months, all stroke patients treated at the Charité Medical Center will be screened retrospectively 9-13 months after a first-ever ischemic stroke (~2000). All eligible patients will be contacted by mail 9-13 months after their hospital stay with the request that they complete the questionnaires. The mailing will also include an information statement, the consent form, as well as a stamped return envelope.

ELIGIBILITY:
Inclusion criteria:

1. Patients treated at the Charité Medical Center for acute ischemic stroke
2. Confirmation of diagnosis by CT or MRI
3. Age > 18 years
4. Ability to give informed consent

Exclusion criteria:

1. Stroke secondary to complications from an intracranial aneurysm, arterial-venous malformation, intracranial tumor or neoplastic process
2. Major diseases at the time of the hospital stay that would be expected to obviate meaningful follow-up assessments such as life-threatening heart or respiratory failure, renal or hepatic failure, cancer

2. Severe comprehension deficits, e.g. severe aphasia, dementia 3. Substantial pre-stroke disability (e.g. from a previous stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the Charité Medical Center for acute ischemic stroke (9-13 months after stroke)
Sampling Method: Probability Sample
Enrollment: 636 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Stroke-induced PTSD | 9-13 months after stroke
  Stroke-induced PTSD will be measured using the Impact of Event Scale - Revised (IES-R).

SECONDARY OUTCOMES:
Trauma exposure | 9-13 months after stroke
  Prior trauma exposure before the infarct is ascertained with the 10-item Brief Trauma Questionnaire (BTQ).
Lifetime PTSD | 9-13 months after stroke
  The occurrence of PTSD symptoms in the study subjects' lifetimes is assessed using the 7-item Short Screening Scale for DSM IV PTSD.
Functional outcome | 9-13 months after stroke
  Functional outcome is measured with the SF-36

OTHER OUTCOMES:
Depression | 9-13 months after stroke
  depressive symptoms are assessed with the BDI (Beck's Depression Inventory)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No